CLINICAL TRIAL: NCT05506371
Title: Azithromycin as an Adjunct to Scaling and Root Planning Causes an Increase of CD68+, CD163+ Macrophages Density in the Gingival Tissues of Periodontitis Patients: a Randomized Controlled Short-term Clinical Trial
Brief Title: Effects of Azithromycin as an Adjunct to Scaling and Root Planning in the Treatment of Periodontitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ukrainian Medical Stomatological Academy (Other)
Responsible Party: Principal Investigator, Igor Kaydashev, Honored Master of Science and Technology of Ukraine, Doctor of Medical Sciences, Professor Vice-Rector for Research and Development of Poltava State Medical University, Ukrainian Medical Stomatological Academy
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0122U00049
Record Dates: First submitted 2022-08-14; First posted 2022-08-18 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Periodontitis
Keywords: Azithromycin; M1 macrophages; M2 macrophages; Macrophages-targeted therapy; Periodontitis
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Intervention Model Description: Randomized controlled short-term clinical trial
Who Masked: Outcomes Assessor
Masking Description: All biopsies were reviewed by the same pathologist, blinded to experimental group affiliation of biopsies
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Az group (Experimental): Periodontitis patients, who underwent scaling and root planning (SRP) as one-stage full-mouth disinfection procedure and additionally received oral azithromycin ("Health" Pharmaceutical Company, Kharkiv, Ukraine) in a dose of 500 mg q.d. for 7 days, then 500 mg q.w. for the next 3 weeks
  Interventions: Drug: Az+SRP
- SRP group (Active Comparator): Periodontitis patients who underwent scaling and root planning (SRP) as one-stage full-mouth disinfection procedure.
  Interventions: Drug: SRP
- H group (Other): Reference group. 25 healthy volunteers who underwent only diagnostics to confirm the clinical healthy state of the gingiva
  Interventions: Drug: No interventions

INTERVENTIONS:
Drug: Az+SRP — Azithromycin as an adjunct to scaling and root planning in the treatment of periodontitis
  Other Names: Azithromicyn group
  Arms: Az group
Drug: SRP — Scaling and root planning (SRP) treatment of periodontitis
  Other Names: Periodontal conventional treatment group
  Arms: SRP group
Drug: No interventions — Diagnostocs to confirm the healthy state of the gingiva
  Other Names: Reference/periodontal health group
  Arms: H group

SUMMARY:
The growing interest in the possibilities of modulating macrophages in inflammatory diseases with therapeutic purpose has prompted the development of new approaches for the treatment of periodontitis.

This randomized add-on open clinical study evaluated the short-term effects of azithromycin (Az) as an adjunct to scaling and root planing (SRP) in patients with chronic periodontitis.

The investigators measured periodontal parameters, and collected gingival biopsies from patients with periodontitis (P group, n=50) before and 1 month after scaling and root planning (SRP group, n=25), after scaling and root planning with oral azithromycin administration (Az group, n=25), and from periodontally healthy individuals (H group, n=25). The last served as a reference group. Macrophage subpopulations were identified through immunohistochemistry as single positive CD68+ and CD163+ cells. The levels of M1-, and M2-related cytokines (IL1-β, IL-6, IL-10, TGF-β) assay in the tissue culture medium was provided by ELISA. The data were statistically analyzed by appropriate methods.

The null hypothesis tested was that L-arginine and L-ornithine have no influences on CD68+ and CD163+ Mφs densities.

DETAILED DESCRIPTION:
Clinical periodontal examinations Periodontal parameters were evaluated at the pre-treatment stage (T0) and 4 weeks ±5 days after the completion of SRP. For all participants, sex and age were recorded, and periodontal parameters such periodontal pocket depth (PPD), clinical attachment loss (CAL), and bleeding on probing (BoP) were examined. All measurements were conducted by one calibrated examiner using a manual periodontal probe (0106.DT06.CP10, Den Tag, Italy). PPD and CAL were measured at six periodontal sites around each tooth (including the third molars) to the nearest 1 mm, and maximal values were taken into account. For H group participants the signs of gingival inflammation, probing depth exceeding 3 mm and BoP were exclude to insure periodontal health.

Periodontal therapy was comprised of home oral hygiene instructions and SRP. It was performed using ultrasonic, Gracey curettes and air-abrasive polishing. Measure for compliance control included counting pills and home hygiene checking.

Collection of gingival tissue samples For precise immunohistochemical study gingival biopsy samples, about 3x3 mm was excised following local anesthesia from all participants without any harm, during appropriate dental procedures. Biopsy from periodontitis-affected gingiva performed at pre-treatment (T0, P Group) and 4 weeks ±5 days after the completion of periodontal treatment, in the same or nearest points, from a single most severe clinical appropriate site around common dental and periodontal procedures such was tooth extraction due to caries complications, and gingivectomies. Biopsy from periodontally healthy patients were obtained during tooth extraction due to caries complications, wisdom teeth and orthodontic indications. After collection, the half of biopsies were fixed in a 4% formalin solution for 24 hours of fixation, dehydrated, and embedded in paraffin, and another half were prepared for cytokines assay.

Immunohistochemistry and antibodies Paraffin sections, 2-3 μm in thickness were deparaffinized and dehydrated. Heat-induced epitope retrieval in citrate buffer, pH 6, was performed by heating the slides in the microwave oven for 23 min, then allowed to cool, rinsed with phosphate-buffered saline (PBS), incubated with blocked reagent, rinsed, and incubated with mouse monoclonal CD68 macrophage antibodies (1:30, clone PG-M1, Diagnostic BioSystems, The Hague, The Netherlands) or anti-CD163 (1:100, clone 10D6, Diagnostic BioSystems, The Hague, The Netherlands). Then sections were stained with the 2-steps plus Mouse/Rabbit PolyVueTM HRP/DAB Detection System (Diagnostic BioSystems, The Hague, The Netherlands), and counterstained with Mayer's haemalaun. PBS was used as negative controls, the lymph node tissue - as a positive control.

Evaluation of immunohistochemical staining СD68+ and CD163+ macrophages were estimated by counting the number of the cells by light microscope in 400 times in intensive cell infiltrative areas, selected 5 regions from each slice, and all 5 counts were taken for further statistics. Immunopositive Mφs in the areas of cell infiltration were count, because of directly relation to the inflammation. The number of cells per 10 000 μm2 was calculated as immunopositive cell density. Photos and calculation were obtained using the light microscope Axio Lab.A1 (Carl Zeiss, Göttingen, Germany) (×400).

Tissue culturing Part of gingival tissue samples were cultured in a humidified incubator at 37 °C and in the presence of 5 % CO2. Biopsies were cultured in Dulbecco's modified Eagle medium (DMEM) supplemented with 10 % (vol/vol) fetal bovine serum (Gibco, Thermo Fisher Scientific, Gibco™, US), 1 % (vol/vol) penicillin-streptomycin (Gibco™, US), and 0.2 % (vol/vol) fungizone amphotericin B (Gibco™, US) during 48 h [16]. For culturing, each biopsy sample was placed in a separate well of Costar® 24-well Plates (Corning Incorporated - Life Sciences, Kennebunk, USA), containing 0,4 ml of supplemented DMEM. After incubation, the tissues were removed and culture media were centrifuged at 800 g and 4 °C.

Cytokine assay Cytokine assay in the tissue culture medium was provided by ELISA. IL1-β, IL-6, IL-10, and TGF-β concentrations were measured by commercially available kits (Vector Best, Novosibirsk, Russia, and MyBioSource, San Diego, USA). Cytokine concentrations were expressed as recommended by the manufacturer.

Statistical analysis Statistical analysis was performed using the Prism 5 software (GraphPad Software, San Diego, USA) by means of nonparametric (descriptive statistics, Wilcoxon matched-pairs signed-rank test - for comparison of dependent results, Mann-Whitney test - for independent groups; nonparametric ANOVA for multiple comparisons with post-hoc tests, and Spearmen correlation). CD68+/CD163+ ratio was assessed by inter-group comparisons and Spearman correlation checking. P values of <0.05 were considered statistically significant in all analyses. For descriptive statistics of cell numbers, the percentile ranges were also used because of non-normal variables distributions.

ELIGIBILITY:
Inclusion criteria for healthy volunteers:

* Presence of more than 20 teeth (for each tooth, the probing pocket depth ≤3 mm
* Absence of clinical gingival inflammation at intact or reduced periodontium

Inclusion Criteria:

* The presence of at least 15 natural teeth, at least 10 sites with the periodontal pocket depth (PPD) ≥4 mm, and/or clinical attachment loss of ≥4 mm at the same site, and satisfactory general health

Exclusion Criteria:

* Taking antibiotics or anti-inflammatory medications within the previous 3 months
* Periodontal therapy within the previous 6 months
* Purulent exudation from periodontal pockets
* Pregnancy or breastfeeding
* Severe, uncontrolled (decompensated) diseases of the internal organs, or neuropsychiatric disorders
* Other conditions that determined the patient's inability to understand the nature and possible consequences of the study

Ages: 19 Years to 54 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2017-09-16 (Actual); Primary Completion 2019-06-28 (Actual); Study Completion 2019-06-28 (Actual)

PRIMARY OUTCOMES:
Change in clinical attachment loss (CAL) | The pre-treatment stage (T0) and 4 weeks ±5 days after the completion of SRP
  Mean CAL, measured at six periodontal sites around each tooth (including the third molars) to the nearest 1 mm
Change in periodontal pocket depth (PPD) | The pre-treatment stage (T0) and 4 weeks ±5 days after the completion of SRP
  Mean periodontal pocket depth, measured at six periodontal sites around each tooth (including the third molars) to the nearest 1 mm

SECONDARY OUTCOMES:
Change in bleeding on probing (BOP) | The pre-treatment stage (T0) and 4 weeks ±5 days after the completion of SRP
  The percentage of sites per patient with bleeding measured at six sites around each tooth (including the third molars)
Change in density of CD68+ macrophages | The pre-treatment stage (T0) and 4 weeks ±5 days after the completion of SRP
  The number of single-immunopositive macrophages per 10 000 μm2 was calculated as cell density in biopsy from periodontitis-affected gingiva
Change in density of CD163+ macrophages | The pre-treatment stage (T0) and 4 weeks ±5 days after the completion of SRP
  The number of single-immunopositive macrophages per 10 000 μm2 was calculated as cell density in biopsy from periodontitis-affected gingiva
Change in mean level of IL1-β in periodontitis-affected gingiva | The pre-treatment stage (T0) and 4 weeks ±5 days after the completion of SRP
  The mean level of IL1-β in the tissue culture medium, obtained from the same biopsy
Change in mean level of IL-6 in periodontitis-affected gingiva | The pre-treatment stage (T0) and 4 weeks ±5 days after the completion of SRP
  The mean level of IL-6 in the tissue culture medium, obtained from the same biopsy
Change in mean level of IL-10 in periodontitis-affected gingiva | The pre-treatment stage (T0) and 4 weeks ±5 days after the completion of SRP
  The mean level of IL-10 in the tissue culture medium, obtained from the biopsy
Change in mean level of TGF-β in periodontitis-affected gingiva | The pre-treatment stage (T0) and 4 weeks ±5 days after the completion of SRP
  The mean level of TGF-β in the tissue culture medium, obtained from the biopsy

CONTACTS AND LOCATIONS:
Overall Officials: Igor P. Kaidashev, MD, Principal Investigator — Ukrainian Medical Stomatological Academy Poltava, Ukraine
Locations (1):
- Department of Postgraduate Education for Dentists of Poltava State Medical University,, Poltava, Ukraine

IPD SHARING:
Plan to Share IPD: No
We plan to provide all the necessary data in a future article.

REFERENCES:
- [Background] Morales A, Contador R, Bravo J, Carvajal P, Silva N, Strauss FJ, Gamonal J. Clinical effects of probiotic or azithromycin as an adjunct to scaling and root planning in the treatment of stage III periodontitis: a pilot randomized controlled clinical trial. BMC Oral Health. 2021 Jan 7;21(1):12. doi: 10.1186/s12903-020-01276-3. PMID 33413320
- [Background] Haffajee AD, Socransky SS, Ebersole JL. Survival analysis of periodontal sites before and after periodontal therapy. J Clin Periodontol. 1985 Aug;12(7):553-67. doi: 10.1111/j.1600-051x.1985.tb01389.x. PMID 3860518
- [Background] Mills CD, Lenz LL, Ley K. Macrophages at the fork in the road to health or disease. Front Immunol. 2015 Feb 16;6:59. doi: 10.3389/fimmu.2015.00059. eCollection 2015. No abstract available. PMID 25762997
- [Background] Zhou LN, Bi CS, Gao LN, An Y, Chen F, Chen FM. Macrophage polarization in human gingival tissue in response to periodontal disease. Oral Dis. 2019 Jan;25(1):265-273. doi: 10.1111/odi.12983. Epub 2018 Oct 12. PMID 30285304
- [Background] Shapouri-Moghaddam A, Mohammadian S, Vazini H, Taghadosi M, Esmaeili SA, Mardani F, Seifi B, Mohammadi A, Afshari JT, Sahebkar A. Macrophage plasticity, polarization, and function in health and disease. J Cell Physiol. 2018 Sep;233(9):6425-6440. doi: 10.1002/jcp.26429. Epub 2018 Mar 1. PMID 29319160
- [Background] Allam JP, Duan Y, Heinemann F, Winter J, Gotz W, Deschner J, Wenghoefer M, Bieber T, Jepsen S, Novak N. IL-23-producing CD68(+) macrophage-like cells predominate within an IL-17-polarized infiltrate in chronic periodontitis lesions. J Clin Periodontol. 2011 Oct;38(10):879-86. doi: 10.1111/j.1600-051X.2011.01752.x. Epub 2011 Aug 31. PMID 21883359
- [Background] Fabriek BO, Dijkstra CD, van den Berg TK. The macrophage scavenger receptor CD163. Immunobiology. 2005;210(2-4):153-60. doi: 10.1016/j.imbio.2005.05.010. PMID 16164022
- [Background] Parnham MJ, Erakovic Haber V, Giamarellos-Bourboulis EJ, Perletti G, Verleden GM, Vos R. Azithromycin: mechanisms of action and their relevance for clinical applications. Pharmacol Ther. 2014 Aug;143(2):225-45. doi: 10.1016/j.pharmthera.2014.03.003. Epub 2014 Mar 11. PMID 24631273
- [Background] Fujise O, Miura M, Hamachi T, Aida Y, Nishimura F. Regenerative effect of azithromycin on periodontitis with different levels of gingival inflammation: three case reports. Aust Dent J. 2014 Jun;59(2):245-51. doi: 10.1111/adj.12177. PMID 24861402
- [Background] Nepokupnaia-Slobodianuk TS, Skripnikov PN. [The clinical effectiveness of long-term azithromycin in patients with chronic generalized periodontitis]. Georgian Med News. 2014 Nov;(236):27-31. Russian. PMID 25541821
- [Background] Hai R, Chu A, Li H, Umamoto S, Rider P, Liu F. Infection of human cytomegalovirus in cultured human gingival tissue. Virol J. 2006 Oct 5;3:84. doi: 10.1186/1743-422X-3-84. PMID 17022821
- [Background] Loos BG, Needleman I. Endpoints of active periodontal therapy. J Clin Periodontol. 2020 Jul;47 Suppl 22(Suppl 22):61-71. doi: 10.1111/jcpe.13253. PMID 31912527
- [Background] Garaicoa-Pazmino C, Fretwurst T, Squarize CH, Berglundh T, Giannobile WV, Larsson L, Castilho RM. Characterization of macrophage polarization in periodontal disease. J Clin Periodontol. 2019 Aug;46(8):830-839. doi: 10.1111/jcpe.13156. Epub 2019 Jun 25. PMID 31152604
- [Background] Zhu L, Zhao Q, Yang T, Ding W, Zhao Y. Cellular metabolism and macrophage functional polarization. Int Rev Immunol. 2015 Jan;34(1):82-100. doi: 10.3109/08830185.2014.969421. Epub 2014 Oct 23. PMID 25340307
- [Background] Zhu LF, Li L, Wang XQ, Pan L, Mei YM, Fu YW, Xu Y. M1 macrophages regulate TLR4/AP1 via paracrine to promote alveolar bone destruction in periodontitis. Oral Dis. 2019 Nov;25(8):1972-1982. doi: 10.1111/odi.13167. Epub 2019 Oct 18. PMID 31361069